CLINICAL TRIAL: NCT06427421
Title: Characterization of Autoreactive Regulatory and Conventional CD4 T Cells in Recent Onset Type 1 Diabetes and Control Individuals
Acronym: CARegT1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP230664; 2024-A00696-41 (Other: ID-RCB)
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Regulatory T cells; Pathophysiology of T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Single-Cell Gene Expression Analysis; Histocompatibility Testing; Glycated Hemoglobin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly diagnosed T1DM group (Other): children aged 2 to under 18 on the day of inclusion, with a recent diagnosis of type 1 diabetes
  Interventions: Biological: Frequency of Treg and Teffs; Biological: Phenotype of Treg and Teffs; Biological: RNA seq analysis; Biological: HLA typing; Biological: beta-cell autoantibody dosage
- Control group (Other): children aged 2 to under 18 on the day of inclusion, with no history of type 1 diabetes
  Interventions: Biological: Frequency of Treg and Teffs; Biological: Phenotype of Treg and Teffs; Biological: RNA seq analysis; Biological: HLA typing; Biological: beta-cell autoantibody dosage; Biological: Glycated haemoglobin (HbA1C) dosage; Biological: blood glucose dosage; Biological: C-peptide dosage

INTERVENTIONS:
Biological: Frequency of Treg and Teffs — additionnal blood sampling at inclusion
Biological: Phenotype of Treg and Teffs — additionnal blood sampling at inclusion
Biological: RNA seq analysis — additionnal blood sampling at inclusion
Biological: HLA typing — additionnal blood sampling at inclusion
Biological: beta-cell autoantibody dosage — additionnal blood sampling at inclusion
Biological: Glycated haemoglobin (HbA1C) dosage — additionnal blood sampling at inclusion
  Arms: Control group
Biological: blood glucose dosage — additionnal blood sampling at inclusion
  Arms: Control group
Biological: C-peptide dosage — additionnal blood sampling at inclusion
  Arms: Control group

SUMMARY:
Type 1 diabetes (T1D) is caused by an autoimmune response leading to the destruction of pancreatic beta cells. The disease association with particular HLA class II alleles, particularly HLA-DQ8, indicates the implication of CD4 T cells in its aetiology. The hypothesis is therefore that T1D starts by the loss of tolerance in autoreactive CD4 T cells. This might result from alterations in conventional autoreactive CD4 T cells (Tcons), which drive disease, or autoreactive regulatory CD4 T cells expressing the transcription factor FOXP3 (Tregs), which normally maintain immune tolerance. The investigators expect that the characterization of HLA-DQ8-restricted Tcons and Tregs in recent onset HLA-DQ8+ T1D patients shall shed light on the molecular mechanisms underpinning T1D development. This knowledge will guide the development of novel cell therapies harnessing the power of genetically engineered Tregs expressing the relevant antigen receptor to restore immune homeostasis upon cell transfer. The ultimate goal is to reach a curative effect

DETAILED DESCRIPTION:
During the development of type 1 diabetes (T1DM), regulatory T cells (Treg) are modified and their protective role is no longer optimal, particularly against pathology-specific autoreactive antigens. The hypothesis is that in patients with T1DM, the function and phenotype of Treg cells, as well as their receptor repertoire for the antigen to which they are specific (TCR), no longer allow them to control tolerance. The in-depth study of these cells, at both genetic and molecular levels, will enable a major breakthrough in our understanding of the pathophysiology of T1DM, and in the development of targeted cell therapy.

The investigators expect major/important differences between patient Tregs and those of the control population in this study, at the molecular, phenotypic and functional levels. These differences will highlight the TCRs recognizing the target self-antigens. In this way, investigators expect to be able to select a limited number of Treg TCRs that could ultimately be used in cell therapy to restore the protective role of Tregs in these patients.

Thus, this knowledge will enable to propose in the future a more effective immunotherapy with a long-term effect, in order to improve the management of patients with autoimmune diabetes and potentially cure them.

Accordingly, yhe investigators will study insulin-specific Tregs in T1DM patients and control individuals, as well as conventional T cells directed against the same antigen, which in patients are implicated in the disease. This will include a study of their functional status, their transcriptomic profile, as well as their TCRs and their fine recognition properties of the major diabetes self-antigen, insulin.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed T1DM group:

* Age ≥ 2 years and < 18 years on day of inclusion;
* Weight ≥ 12 kg;
* Newly diagnosed T1DM, diagnosis defined according to International Society of Pediatric and Adolescent Diabetes (ISPAD) criteria by: hyperglycemia > 2g/L and/or ketonemia and/or polyuro-polydipsia and/or weight loss ;
* Absence of other associated inflammatory or autoimmune diseases;
* Affiliation with a health insurance scheme or beneficiary (excluding AME);
* Written consent of parental guardians;
* Ability to understand and read French.

Control group :

* Age ≥ 2 years and < 18 years on the day of inclusion;
* Weight ≥ 12 kg;
* No personal history of T1DM;
* Affiliation with a health insurance scheme or entitled person (excluding AME);
* Written consent from parental guardians;
* Ability to understand and read French.

Exclusion Criteria:

Newly diagnosed T1DM group:

* Use of oral or intravenous corticosteriods in the month prior to blood sampling
* Contraindication to the use of anaesthetic cream for blood sampling.

Control group :

* History of autoimmune or inflammatory disease
* Use of oral or intravenous corticosteriods in the month prior to blood sampling
* Contraindication to the use of anaesthetic cream for blood sampling

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Frequency and phenotype of Tregs | Within 4 weeks of T1DM diagnosis
  study the frequency and phenotype of insulin-specific autoreactive Tregs lymphocytes among CD4+ T lymphocytes in children with T1DM and compare these values with those of controls. These parameters will be analyzed by flow cytometry using immune cells from blood samples taken from the T1DM and control groups.

SECONDARY OUTCOMES:
HLA testing | Within 4 weeks of T1DM diagnosis
  Description : the HLA of T1DM and controls will be analyzed by qPCR. This will make it possible to associate the results obtained during the analysis of the main criteria with the HLA of each individual.
Isolate insulin-specific Tregs and Teffs cells | Within 4 weeks of T1DM diagnosis
  Insulin-specific Tregs and Teffs cells will be isolated by flow cytometry
Treg and Teffs transcriptome | Within 4 weeks of T1DM diagnosis
  their transcriptome and TCR will be determined by single-cell transcriptomics analysis (scRNAseq).
Full TCR repertoire of Tregs and Teffs | Within 4 weeks of T1DM diagnosis
  Following flow cytometry, the different repertoires will be compared between the DT1 and control groups.
Machine learning analysis | Within 4 weeks of T1DM diagnosis
  Machine learning analysis of the data obtained (TCR, transcriptome, frequency and phenotype of insulin-specific Tregs and Teffs) to predict the relationship between TCR and functional properties of Tregs and Teffs in patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Simon FILATREAU, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patterson CC, Harjutsalo V, Rosenbauer J, Neu A, Cinek O, Skrivarhaug T, Rami-Merhar B, Soltesz G, Svensson J, Parslow RC, Castell C, Schoenle EJ, Bingley PJ, Dahlquist G, Jarosz-Chobot PK, Marciulionyte D, Roche EF, Rothe U, Bratina N, Ionescu-Tirgoviste C, Weets I, Kocova M, Cherubini V, Rojnic Putarek N, deBeaufort CE, Samardzic M, Green A. Trends and cyclical variation in the incidence of childhood type 1 diabetes in 26 European centres in the 25 year period 1989-2013: a multicentre prospective registration study. Diabetologia. 2019 Mar;62(3):408-417. doi: 10.1007/s00125-018-4763-3. Epub 2018 Nov 28. PMID 30483858
- [Background] Mobasseri M, Shirmohammadi M, Amiri T, Vahed N, Hosseini Fard H, Ghojazadeh M. Prevalence and incidence of type 1 diabetes in the world: a systematic review and meta-analysis. Health Promot Perspect. 2020 Mar 30;10(2):98-115. doi: 10.34172/hpp.2020.18. eCollection 2020. PMID 32296622
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Bougneres PF, Carel JC, Castano L, Boitard C, Gardin JP, Landais P, Hors J, Mihatsch MJ, Paillard M, Chaussain JL, et al. Factors associated with early remission of type I diabetes in children treated with cyclosporine. N Engl J Med. 1988 Mar 17;318(11):663-70. doi: 10.1056/NEJM198803173181103. PMID 3125434
- [Background] Parving HH, Tarnow L, Nielsen FS, Rossing P, Mandrup-Poulsen T, Osterby R, Nerup J. Cyclosporine nephrotoxicity in type 1 diabetic patients. A 7-year follow-up study. Diabetes Care. 1999 Mar;22(3):478-83. doi: 10.2337/diacare.22.3.478. PMID 10097932
- [Background] Herold KC, Bundy BN, Long SA, Bluestone JA, DiMeglio LA, Dufort MJ, Gitelman SE, Gottlieb PA, Krischer JP, Linsley PS, Marks JB, Moore W, Moran A, Rodriguez H, Russell WE, Schatz D, Skyler JS, Tsalikian E, Wherrett DK, Ziegler AG, Greenbaum CJ; Type 1 Diabetes TrialNet Study Group. An Anti-CD3 Antibody, Teplizumab, in Relatives at Risk for Type 1 Diabetes. N Engl J Med. 2019 Aug 15;381(7):603-613. doi: 10.1056/NEJMoa1902226. Epub 2019 Jun 9. PMID 31180194
- [Background] Keymeulen B, Vandemeulebroucke E, Ziegler AG, Mathieu C, Kaufman L, Hale G, Gorus F, Goldman M, Walter M, Candon S, Schandene L, Crenier L, De Block C, Seigneurin JM, De Pauw P, Pierard D, Weets I, Rebello P, Bird P, Berrie E, Frewin M, Waldmann H, Bach JF, Pipeleers D, Chatenoud L. Insulin needs after CD3-antibody therapy in new-onset type 1 diabetes. N Engl J Med. 2005 Jun 23;352(25):2598-608. doi: 10.1056/NEJMoa043980. PMID 15972866
- [Background] Vignali DA, Collison LW, Workman CJ. How regulatory T cells work. Nat Rev Immunol. 2008 Jul;8(7):523-32. doi: 10.1038/nri2343. PMID 18566595
- [Background] Corthay A. How do regulatory T cells work? Scand J Immunol. 2009 Oct;70(4):326-36. doi: 10.1111/j.1365-3083.2009.02308.x. PMID 19751267
- [Background] Visperas A, Vignali DA. Are Regulatory T Cells Defective in Type 1 Diabetes and Can We Fix Them? J Immunol. 2016 Nov 15;197(10):3762-3770. doi: 10.4049/jimmunol.1601118. PMID 27815439
- [Background] Bluestone JA, Buckner JH, Fitch M, Gitelman SE, Gupta S, Hellerstein MK, Herold KC, Lares A, Lee MR, Li K, Liu W, Long SA, Masiello LM, Nguyen V, Putnam AL, Rieck M, Sayre PH, Tang Q. Type 1 diabetes immunotherapy using polyclonal regulatory T cells. Sci Transl Med. 2015 Nov 25;7(315):315ra189. doi: 10.1126/scitranslmed.aad4134. PMID 26606968
- [Background] Marek-Trzonkowska N, Mysliwiec M, Dobyszuk A, Grabowska M, Techmanska I, Juscinska J, Wujtewicz MA, Witkowski P, Mlynarski W, Balcerska A, Mysliwska J, Trzonkowski P. Administration of CD4+CD25highCD127- regulatory T cells preserves beta-cell function in type 1 diabetes in children. Diabetes Care. 2012 Sep;35(9):1817-20. doi: 10.2337/dc12-0038. Epub 2012 Jun 20. PMID 22723342
- [Background] Dong S, Hiam-Galvez KJ, Mowery CT, Herold KC, Gitelman SE, Esensten JH, Liu W, Lares AP, Leinbach AS, Lee M, Nguyen V, Tamaki SJ, Tamaki W, Tamaki CM, Mehdizadeh M, Putnam AL, Spitzer MH, Ye CJ, Tang Q, Bluestone JA. The effect of low-dose IL-2 and Treg adoptive cell therapy in patients with type 1 diabetes. JCI Insight. 2021 Sep 22;6(18):e147474. doi: 10.1172/jci.insight.147474. PMID 34324441
- [Background] Kieback E, Hilgenberg E, Stervbo U, Lampropoulou V, Shen P, Bunse M, Jaimes Y, Boudinot P, Radbruch A, Klemm U, Kuhl AA, Liblau R, Hoevelmeyer N, Anderton SM, Uckert W, Fillatreau S. Thymus-Derived Regulatory T Cells Are Positively Selected on Natural Self-Antigen through Cognate Interactions of High Functional Avidity. Immunity. 2016 May 17;44(5):1114-26. doi: 10.1016/j.immuni.2016.04.018. PMID 27192577
- [Background] Krischer JP; Type 1 Diabetes TrialNet Study Group. The use of intermediate endpoints in the design of type 1 diabetes prevention trials. Diabetologia. 2013 Sep;56(9):1919-24. doi: 10.1007/s00125-013-2960-7. Epub 2013 Jun 7. PMID 23744306
- [Background] Noble JA. Immunogenetics of type 1 diabetes: A comprehensive review. J Autoimmun. 2015 Nov;64:101-12. doi: 10.1016/j.jaut.2015.07.014. Epub 2015 Aug 10. PMID 26272854
- [Background] Caillat-Zucman S, Garchon HJ, Timsit J, Assan R, Boitard C, Djilali-Saiah I, Bougneres P, Bach JF. Age-dependent HLA genetic heterogeneity of type 1 insulin-dependent diabetes mellitus. J Clin Invest. 1992 Dec;90(6):2242-50. doi: 10.1172/JCI116110. PMID 1469084
- See also: Related Info — https://diabetesatlas.org/data/